CLINICAL TRIAL: NCT02360722
Title: Improving Nutritional Status With Oral Nutritional Supplement in Chinese Elderly
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was cancelled due to change in food registration regulations in China.
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BL26
Record Dates: First submitted 2015-01-27; First posted 2015-02-11 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-11

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition | interventions — Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral Nutritional Supplement (Experimental): ONS + Nutritional education
  Interventions: Other: Oral Nutritional Supplement; Other: Nutritional Education
- Control Group (Other): Nutritional education only
  Interventions: Other: Nutritional Education

INTERVENTIONS:
Other: Oral Nutritional Supplement — Will receive ONS twice a day for 6 months and two nutritional education at baseline and 3 months after intervention
  Arms: Oral Nutritional Supplement
Other: Nutritional Education — Two nutritional education courses at baseline and 3 months after intervention

SUMMARY:
This is a single- country, interventional, double-arm study involving Chinese Elderly subjects.

DETAILED DESCRIPTION:
This study aims to understand the following:

1. The effect of long-term Oral Nutritional Supplementation (ONS) on improving nutritional and health status in Chinese elderly.
2. The impact of long-term ONS on health cost including both medical cost and social health care burdens.
3. The impact of long-term ONS on life quality of the elderly. The study includes Screening Visit (Day -7~0), and Visit 1(Day 0) to Visit 7 (Day 168±3). Enrollment of anticipated 666 subjects, Male or female Chinese ages >= 60 years, to get 400 evaluable subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female Chinese ages >= 60 years.
2. Subject is ambulatory.
3. Subject with risks of malnutrition defined as DETERMINE score >=3
4. Subject's BMI is below 28.
5. Subject has experienced hospital stay or surgery within 6 months prior to enrollment;
6. Subject if takes any medications for concomitant chronic diseases should be in stable dosage for at least 3 weeks.
7. Subject plans to live in the community for more than 6 months after recruitment.
8. Subject has voluntarily signed and dated an informed consent form, approved by an Independent Ethics Committee/Institutional Review Board (IEC/IRB) prior to any participation in the study.

Exclusion Criteria:

1. Subject has history of allergy to any ingredient in the study product
2. Subject dislikes the experimental product
3. Subject has been diagnosed with diabetes.
4. Subject who has malignancy expected to receive chemotherapy/ radiotherapy scheduled during the study period,
5. Subject has a life expectancy less than 6 months.
6. Subject who has reported chronic liver disease or liver cirrhosis or liver failure or any liver diseases not suitable for the study as the study physician's opinion.
7. Subject who has reported impacted renal function as eGFR < 30 mL/min/1.73 m2 or renal dysfunction severe greater than stage 4 or any other renal diseases not suitable for the study as the study physician' s opinion.
8. Subject who has experienced fever or diarrhea within one week prior to enrollment.
9. Subject who is expected to have scheduled major surgery during the study period.
10. Subject who has physical disabilities such as loss of hand or foot or limbs or any other physical disability which may affect the muscle mass measurement by the opinion of the study physician.
11. Subject has an implanted electronic device or orthopedic metal implantations, such as pacemaker, cardiac defibrillator, subcutaneous injection pump, or metal hip, metal knee joint, metal fracture internal fixation, etc.
12. Subject who has active tuberculosis (TB), hepatitis, or HIV infection as self-reported at enrollment.
13. Subject has severe dementia or delirium, brain metastases, eating disorder, history of significant neurological or psychiatric disorder, or other conditions that may interfere with study product consumption or compliance with study protocol procedures in the opinion of the principal investigator or study physician.
14. Subject is drug addicted or alcohol addicted
15. Subject has any other disease or situation who should not to participate in the study by the opinion of study physicians.
16. Subject is participating in other clinical trials which are not approved by AN

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-10; Primary Completion 2017-07 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change of body weight from baseline to the end of the study | 24 weeks

SECONDARY OUTCOMES:
Total number of sick days due to Upper Respiratory Tract Infections (URTI) | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xianfeng ZHAO, MD, PhD, Study Chair — Abbott Nutrition R&D China

IPD SHARING:
Plan to Share IPD: No